CLINICAL TRIAL: NCT00584636
Title: Nebulized Budesonide After Discharge From a Pediatric Emergency Department in Preventing Asthma Relapse: A Randomized, Double-Blind, Placebo Controlled Trial.
Brief Title: Pulmicort Respules on Relapse Rates After Treatment in the ED
Acronym: Budesonide
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study halted prematurely before enrollment of first patient
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRUSBUPR0034
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2011-09

CONDITIONS: Asthma
Keywords: child; emergency department
MeSH Terms: conditions — Asthma; Emergencies | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pulmicort Respules (Experimental): using pulmicort respules
  Interventions: Drug: pulmicort respules

INTERVENTIONS:
Drug: pulmicort respules — pulmicort respules 0.5 mg twice a day for 28 days versus placebo
  Other Names: Budesonide

SUMMARY:
The purpose of this study is to see if the addition of budesonide to oral corticosteroids will result in a decrease in relapse rates compared to oral corticosteroids alone in children who are discharged from the ED after an asthma exacerbation. Secondly, that there will be an improvement in lung function, a decrease in beta-2 agonist use and an improvement in health-related quality of life compared to placebo.

DETAILED DESCRIPTION:
Children between the ages of 2 and 8 years inclusive who have a history of asthma are eligible for enrollment if they present to the pediatric emergency department with an asthma exacerbation that is believed would not require admission to the hospital. All eligible children will be enrolled whenever there are study personnel available after obtaining informed written consent. Children less than 2 years of age will not be enrolled as their wheezing may be due to bronchiolitis. Children will also be excluded if they have been on an oral or inhaled corticosteroid in the last week, have a history of a chronic lung disease (e.g. cystic fibrosis), non-corrected congenital heart disease, are pregnant, or unavailable for follow-up.

Initial asthma severity will be based on PEFR's or clinical asthma scores (table 1). If the child is able to reliably provide a peak flow in the emergency department this value will be recorded and calculated as a percentage of their predicted based on standardized height and weight charts. All peak flows will be performed by licensed respiratory therapists or trained registered nurses. If a childs effort during the performance of the peak flows is considered poor by the respiratory therapist then only the asthma score will be utilized. If a child can perform the peak flows adequately they will be sent home with the peak flow meter. All children will be assigned clinical asthma scores regardless of whether peak flows are obtained. With this asthma scale a score of less than 7 is considered mild, 8 to 11 moderate and a score of 12 to 15 severe. This asthma score has been shown to have good interobserver reliability with a Pearson correlation statistic of 0.92.

Children will be treated based on normal practice patterns for our ED and the decision to discharge a patient will be at the attending physician's discretion. All children will receive 2 mg/kg of methylprednisolone up to a maximum dose of 60 mg orally within the first 60 minutes of treatment or 0.6mg/kg of oral dexamethasone (max 15mg) given in the Emergency room. When discharged home all children will be given a prescription for 4 days of methylprednisolone in a dose of 1 mg/kg given once daily Patients will be assigned in a double blind fashion to budesonide nebules or placebo. A computer generated table of random numbers will be used to assign children to treatment group. Groups will be randomized in blocks of 10. A locked area in the ED will contain numbered plastic bags each containing either budesonide nebules or identical appearing and tasting placebo nebules. Study personnel and patients will be blinded to treatment allocation for the entire length of the trial. Patients will be given instructions on the use and dosage (based on weight) of the study medications.

All patients will be contacted by telephone at 7 days. They will be followed for 28 days or until they relapse, whichever comes first. Relapse will be defined as any unscheduled physician visit for worsening asthma symptoms. At the time of telephone follow-up patients will be asked about symptoms as well as about compliance with their study medications (see data collection sheet). At the return visit on day 28 they will be asked to bring their medication with them to determine compliance. At that time they will also have peak flows obtained and a repeat assessment of the quality of life scale.

In order to measure health-related quality of life, the Integrated Therapeutics Group Child Asthma Short Form (ITG-CASF) will be completed by a research assistant upon enrollment, via telephone follow-up 7 days after the emergency department visit, and at the 28 day follow-up visit. The ITG-CASF has previously been validated in children with chronic asthma. Gorelick et al have shown it to be a valid and responsive measure of health-related quality of life in children as young as 2 years of age treated in an emergency department for acute asthma. The 8-item ITG Child Asthma Short Form measures the following three concepts: Daytime Symptoms, Nighttime Symptoms, and Functional Limitations. In addition to the standard 8-item ITG Child Asthma Short Form, they identified two additional items from the long form to assess whether inhaler use interfered with the child's life and whether adjustments were made to family life because of the child's asthma.

ELIGIBILITY:
Inclusion Criteria:

Patient is between the ages of 2 and 8

* Has previously been diagnosed with asthma by any physician
* Has presented to the ED with an asthma exacerbation judged by a physician that is believed would not required admission to the hospital

Exclusion Criteria:

* Children less than 2 years (wheezing may be due to bronchiolitis)
* Children who have been on oral or inhaled corticosteroid in the last week, are pregnant, or unavailable for follow-up
* Pregnant
* Has chronic lung diseases (i.e. cystic fibrosis)

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of unplanned ED or PCP visits for asthma in the 1 month following an ED visit for an asthma exacerbation. | 28 days

SECONDARY OUTCOMES:
Use of rescue medications, hospitalizations and quality of life questionaires. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Bulloch, MD, Principal Investigator — Phoenix Children's Hospital; Katherine Mandeville, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States